CLINICAL TRIAL: NCT06454669
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Groups Study to Explore the Safety and Therapeutic Potential of Dronabinol as an Adjunct for Reducing Pain
Brief Title: Dronabinol as an Adjunct for Reducing Pain
Acronym: DARP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher D. Verrico (Other)
Responsible Party: Sponsor-Investigator, Christopher D. Verrico, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-51389
Record Dates: First submitted 2024-04-18; First posted 2024-06-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain; Chronic Pain; Back Injuries
Keywords: dronabinol; Marinol; THC
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Injuries | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel Groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Dronabinol (Experimental): Dronabinol capsules, over-encapsulated with filler to match the appearance of the placebo capsule, up to 15 mg, twice per day for 8 weeks.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Capsules with placebo (i.e., cellulose filler), twice per day for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Eligible subjects will be randomized (2:1) to dronabinol or placebo, administered orally. The dose of dronabinol will be titrated such that on Day 1, subjects will take 2.5 mg, twice. On subsequent days patients may gradually increase the total number of doses, by one dose each day, as needed and tolerated until either the optimal dose is achieved, or the dose reaches 30 mg THC per day.
  Other Names: Marinol; delta-9-tetrahydrocannabinol
  Arms: Drug: Dronabinol
Drug: Placebo — Matching placebo will be prepared and administered in the same manner as the active medication. Titration will occur in a masked fashion such that individuals assigned to placebo undergo a similar perceived titration process.
  Arms: Placebo

SUMMARY:
This exploratory, proof-of-concept study is a double-blind (participants and investigators will be blinded), placebo-controlled, randomized, two-arm clinical trial of Marinol [dronabinol, synthetic Δ9-tetrahydrocannabinol (THC)] for chronic low back pain (cLBP) with a 2:1 allocation ratio. Up to 75 subjects will be enrolled in this pilot study and randomized to receive doses of THC (up to 30 mg/day), orally, over 8 weeks. This study will be conducted at a single site; it does not include any stratifications, and there is no interim analysis planned. Notably, the goal is to determine whether there is enough evidence of the safety of THC to support the development of later-phase clinical trials. Thus, detailed developmental plans are contingent on the outcomes of this study.

DETAILED DESCRIPTION:
Musculoskeletal pain can be due to an injury to the bones, joints, muscles, tendons, ligaments, or nerves, which can be caused by jerking movements, car accidents, falls, fractures, sprains, dislocations, and direct blows to the muscle. Musculoskeletal pain can be localized in one area, or widespread. Lower back pain is the most common type of musculoskeletal pain. Other common types include tendonitis, myalgia (muscle pain), and stress fractures. A review of opioids for non-cancer musculoskeletal diseases concluded that opioids were "only slightly more effective than their placebos, no more effective than acetaminophen, and somewhat less effective than nonsteroidal anti-inflammatory drugs. In fact, the Centers for Disease Control (CDC) recommends that opioids should not be considered an option for chronic musculoskeletal pain. The impact of cannabinoid treatments on pain in human volunteers has been evaluated for: 1) experimentally induced acute pain, 2) acute postsurgical pain, and 3) chronic pain. Collectively, these data suggest that cannabinoids may be more effective for chronic rather than acute pain conditions. However, there have been few randomized, double-blind, placebo-controlled clinical trials (RCTs, the "Gold Standard" in intervention-based studies) of cannabinoids for pain. To this end, the proposed study will contribute to the evidence base concerning the potential utility of treating chronic low back pain (cLBP) with cannabinoids.

Four RCTs in 159 patients with fibromyalgia, osteoarthritis, chronic back pain, and rheumatoid arthritis treated with oral cannabinoids (nabilone, THC/cannabidiol (CBD), and fatty acid amide hydrolase (FAAH) inhibitor, placebo, or active control (amitriptyline), were included in a systemic review. The results were inconsistent and did not reveal whether the cannabinoids were superior to the controls (placebo and amitriptyline). The authors concluded that there is insufficient evidence for the recommendation for cannabinoid use for pain management in patients with rheumatic diseases. Since then, a Phase II RCT (65 participants) found no difference between THC and placebo in reducing pain measures in patients with chronic abdominal pain due to surgery or chronic pancreatitis.

A more recent systematic review and meta-analysis aimed to "analyze the evidence surrounding the benefits and harms of medical cannabinoids in the treatment of chronic, non-cancer-related pain". Thirty-six trials (4006 participants) were included, examining smoked cannabis (4 trials), oromucosal cannabis sprays (14 trials), and oral cannabinoids (18 trials). Of the 18 trials that examined oral cannabinoids, 15 examined synthetic THC in the form of dronabinol (n=9), nabilone (n=4), or nasimol (n=2). Treatment durations ranged from 1 day to 6 months. Across the 29 trials (34 comparisons) that had reported on pain outcomes, there was a significant treatment effect favoring the use of cannabinoids over placebo (-0.63, 95% confidence interval (CI), -0.85 to -0.42, I2 = 16%, P < 0.00001). Compared with placebo, cannabinoids showed a significant reduction in pain, which was greatest with treatment duration of 2 to 8 weeks (weighted mean difference on a 0-10 pain visual analog scale -0.68, 95% CI, -0.96 to -0.40, I2 = 8%, P < 0.00001; n = 16 trials). Across all time points, oral formulations demonstrated a superior effect compared with oromucosal and inhaled routes of administration. Serious AEs were rare, and similar across the cannabinoid (74 out of 2176, 3.4%) and placebo groups (53 out of 1640, 3.2%). There was an increased risk of non-serious adverse events (AEs) with cannabinoids compared with placebo. Overall, the authors found that cannabinoids are an effective form of pain control in this patient population, with a particularly strong effect among those cannabinoids that are orally administered. However, these studies were found to be limited by overall quality, which were largely underpowered, selective, and inconsistent in their reporting. This preliminary evidence of effectiveness indicates the need for high-quality RCTs in orthopedic areas.

The FDA has not approved a cannabinoid medication to treat cLBP. Here the investigators propose to study the effects of THC for several reasons. First, although both smoked cannabis and THC decrease pain sensitivity, increase pain tolerance, and decrease subjective ratings of pain intensity, THC produces more consistent analgesia for a longer duration. Second, the therapeutic effects of cannabinoids are best established for THC. Third, defined substances, such as purified cannabinoid compounds, are preferable to plant products, which are of variable and uncertain composition. Use of defined cannabinoids permits a more precise evaluation of their effects, whether combined or alone. Finally, compared with marijuana, THC produces lower ratings of abuse-related subjective effects, which can be predictive of use and abuse patterns. Hence, the investigators have elected to study THC. The primary objective of this double-blind, randomized, placebo-controlled, 1-site study is to explore the safety and tolerability of THC, versus placebo when orally administered to patients suffering from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Ability to take oral medication per protocol.
4. Male or female, aged 18-64 years.
5. Has chronic low back pain (i.e., in the space between the lower posterior margin of the rib cage and the horizontal gluteal fold) that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months (Items 1 & 2 from the Research Standards for Chronic Low-Back Pain (RScLBP) assessment).
6. For females of reproductive potential: currently practicing an effective form of two types of birth control, which are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, for at least 1 month prior to screening and agrees to use such a method during study participation and for an additional 4 weeks after the end of study medication administration unless she is surgically sterile, partner is surgically sterile, or she is postmenopausal (one year):

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. etonogestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. complete abstinence from sexual intercourse, and/or hormonal vaginal contraceptive ring.
7. Agree (if male) to use acceptable methods of contraception if the male participant's partner could become pregnant from the time of the first administration of the study drug until 30 days following the final administration of the study drug. One of the following acceptable methods of contraception must be utilized:

   1. Surgical sterilization (vasectomy)
   2. The participant's female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or sub dermal implants (commenced at least 14 days prior to study drug administration to the male participant)
   3. The participant's female partner uses a medically prescribed topically applied transdermal contraceptive patch (commenced at least 14 days prior to study drug administration to the male participant)
   4. The participant's female partner has undergone tubal ligation (female sterilization) or is postmenopausal (one year)
   5. The participant's female partner has undergone placement of an intrauterine device or intrauterine system.
   6. True abstinence: when this is in line with the preferred and usual lifestyle of the participant.
8. Agreement to adhere to Lifestyle Considerations throughout study duration.
9. On a stable pain treatment (pharmacological or otherwise) for ≥3 months at the time of the screening.

Exclusion Criteria:

1. Current and unwilling to stop use of cannabis/marijuana and any other cannabinoids, including over the counter CBD products.
2. Known allergic reactions to cannabis, CBD, THC, or components of the study interventions.
3. Have Blood Urea Nitrogen or Creatinine levels outside the normal range, or other clinically significant laboratory abnormalities.
4. Current use of Antiepileptic drugs.
5. Current use of barbiturates, benzodiazepines, ethanol, lithium, buspirone, muscle relaxants
6. Current use of amphetamines, other sympathomimetic agents, atropine, amoxapine, scopolamine, antihistamines, other anticholinergic agents, amitriptyline, desipramine, or other tricyclic antidepressants within 3 months of randomization.
7. Treatment with another investigational drug or other intervention within 3 months of the screening visit.
8. Pregnancy, plans to become pregnant, or lactation.
9. Any interventional pain procedures within 6 weeks prior to screening or at any point during study enrollment.
10. Surgical intervention or introduction/increased dose of an opioid or analgesic regimen at any point during study enrollment.
11. Implanted spinal cord or dorsal root ganglion stimulator for pain treatment.
12. Meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for a current major psychiatric illness, such as bipolar disorder, major depression, or psychosis.
13. Have a history of substance abuse or dependence.
14. Have a history or current suicidality. Have an increased risk of suicide that necessitates inpatient treatment or warrants therapy excluded by the protocol, and/or current suicidal plan, per investigator clinical judgement, based on interview and defined on the Columbia Suicidality Severity Rating Scale (C-SSRS).
15. Have a history of seizures.
16. Have uncontrolled renal, hepatic, or other systemic disorders that in the opinion of the investigator may jeopardize the patient.
17. Have a history of cardiac disorders.
18. Myocardial infarction or stroke in the previous 6 months.
19. Resting heart rate of > 120.
20. Systolic blood pressure > 140 mm Hg, or diastolic blood pressure > 90 mm Hg.
21. Any uncontrolled communicable disease (e.g., human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), tuberculosis, coronavirus disease (COVID), etc.).
22. Have any other illness, condition, or use of medications, which in the opinion of the P.I. and/or the admitting clinician would preclude the safe and/or successful completion of the study.
23. Have a history of head trauma, epilepsy, or a cognitive disorder (Alzheimer's Disease, dementia).
24. Have an electrocardiogram (ECG) abnormalities at screening including but not limited to bradycardia (<55 beats per minute); prolonged heart-rate corrected QT interval (QTc) interval (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block; pre-existing severe gastrointestinal narrowing (pathologic or iatrogenic).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline to 8-weeks
  For change in pain intensity from baseline to 8-weeks, the investigators will estimate the mean within each arm using the Research Standards for Chronic Low-Back Pain (RScLBP).
Safety Analysis - Adverse Events (AEs) | Baseline to 8-weeks
  AEs will be coded using the most recent version of the Medical Dictionary of Regulatory Activities (MedDRA) preferred terms and will be grouped by system, organ, and class (SOC) designation. The severity, frequency, and relationship of AEs to investigational product will be presented by preferred term by SOC grouping. Listings of each individual AE including start date, stop date, severity, relationship, outcome, and duration will be provided.

SECONDARY OUTCOMES:
Analgesic Use Log | Baseline to 8-weeks
  Analgesic Use Change in Analgesic Use Log scores Day 1 to 56 Secondary analyses will use proper tests and appropriate statistical methods at a significance level of 0.05 (2-sided).
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | Baseline to 8-weeks
  The severity of pain will be assessed by the validated scale within the Patient-Reported Outcomes Measurement Information System (PROMIS).
Profile of Mood States (POMS questionnaire) | Baseline to 8-weeks
  Changes in POMS . Scale range is 1 to 5 and describes how you feel right now. Scale of 1, the lowest score, describes a feeling of Not At All right now for the mood and the scale of 5 gives the highest score representing a feeling of Extremely for the mood.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Verrico, phD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E Debakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Fitzcharles MA, Baerwald C, Ablin J, Hauser W. Efficacy, tolerability and safety of cannabinoids in chronic pain associated with rheumatic diseases (fibromyalgia syndrome, back pain, osteoarthritis, rheumatoid arthritis): A systematic review of randomized controlled trials. Schmerz. 2016 Feb;30(1):47-61. doi: 10.1007/s00482-015-0084-3. PMID 26767993
- [Background] Johal H, Devji T, Chang Y, Simone J, Vannabouathong C, Bhandari M. Cannabinoids in Chronic Non-Cancer Pain: A Systematic Review and Meta-Analysis. Clin Med Insights Arthritis Musculoskelet Disord. 2020 Feb 19;13:1179544120906461. doi: 10.1177/1179544120906461. eCollection 2020. PMID 32127750
- [Background] Kraft B, Frickey NA, Kaufmann RM, Reif M, Frey R, Gustorff B, Kress HG. Lack of analgesia by oral standardized cannabis extract on acute inflammatory pain and hyperalgesia in volunteers. Anesthesiology. 2008 Jul;109(1):101-10. doi: 10.1097/ALN.0b013e31817881e1. PMID 18580179
- [Background] Madden A. Commentary on Madden et al. (2018): 'It's not only about the destination... it's also about the journey!' Consumer perspectives on a model of open-access MAT provision. Addiction. 2018 Aug;113(8):1459-1460. doi: 10.1111/add.14273. No abstract available. PMID 29998623
- [Background] Cooper C, Spiers N, Livingston G, Jenkins R, Meltzer H, Brugha T, McManus S, Weich S, Bebbington P. Ethnic inequalities in the use of health services for common mental disorders in England. Soc Psychiatry Psychiatr Epidemiol. 2013 May;48(5):685-92. doi: 10.1007/s00127-012-0565-y. Epub 2012 Aug 15. PMID 22893107
- [Background] Berthelot JM, Darrieutort-Lafitte C, Le Goff B, Maugars Y. Strong opioids for noncancer pain due to musculoskeletal diseases: Not more effective than acetaminophen or NSAIDs. Joint Bone Spine. 2015 Dec;82(6):397-401. doi: 10.1016/j.jbspin.2015.08.003. Epub 2015 Oct 6. PMID 26453108
- [Background] de Vries JD, van Hooff MLM, Geurts SAE, Kompier MAJ. Exercise to reduce work-related fatigue among employees: a randomized controlled trial. Scand J Work Environ Health. 2017 Jul 1;43(4):337-349. doi: 10.5271/sjweh.3634. Epub 2017 Mar 21. PMID 28323305